CLINICAL TRIAL: NCT05361668
Title: A Randomized, Parallel Group Study to Evaluate the Safety, Pharmacokinetics, and Dose Response of Paltusotine Treatment in Subjects With Carcinoid Syndrome
Brief Title: Study to Evaluate the Safety, PK, and Dose Response of Paltusotine in Subjects With Carcinoid Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRN00808-11
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Carcinoid Syndrome; Carcinoid; Carcinoid Tumor; Carcinoid Tumor of Ileum; Carcinoid Tumor of Cecum; Carcinoid Syndrome Diarrhea; Carcinoid Intestine Tumor; Carcinoid Tumor of Liver; Carcinoid Tumor of Pancreas
Keywords: Neuroendocrine tumor; Paltusotine; CRN00808; Carcinoid syndrome; Lanreotide; Octreotide; Somatostatin agonist
MeSH Terms: conditions — Serotonin Syndrome; Carcinoid Tumor; Carcinoid Tumors, Intestinal; Neuroendocrine Tumors | interventions — Random Allocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 40 mg Paltusotine (Experimental): Participants received paltusotine 40mg, in tablet form, orally, daily, for 8 weeks.
  Interventions: Drug: Randomized: 40 mg Paltusotine
- 80 mg Paltusotine (Experimental): Participants received paltusotine 80mg, in tablet form, orally, daily for 8 weeks.
  Interventions: Drug: Randomized: 80 mg Paltusotine

INTERVENTIONS:
Drug: Randomized: 40 mg Paltusotine — Two 20 mg tablets QD (Potential post-randomization dose escalation based on efficacy and acceptable tolerability: up to 80 mg)
  Arms: 40 mg Paltusotine
Drug: Randomized: 80 mg Paltusotine — Four 20 mg tablets QD (Potential post-randomization dose escalation based on efficacy and acceptable tolerability: up to 120 mg)
  Arms: 80 mg Paltusotine

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), and exploratory dose response of paltusotine treatment in subjects with carcinoid syndrome. This study consists of a Randomized Treatment Phase followed by an Open-Label Extension (OLE) Phase.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, open-label, parallel-group, multicenter study designed to evaluate the safety, pharmacokinetics, and efficacy of paltusotine treatment in subjects with carcinoid syndrome. The study was conducted in 2 parts: a Randomized Treatment Phase (RTP) which is completed, and an Open-label Extension (OLE) Phase which is still ongoing. The RTP consisted of paltusotine treatment for 8 weeks. Subjects who completed the RTP were eligible to enter the OLE Phase at the recommendation of the Investigator. In the ongoing OLE Phase, paltusotine is being administered for a further 102 weeks. The total duration of paltusotine treatment for the combined RTP and OLE Phase is up to 110 weeks (28 months).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age. 2. Documented carcinoid syndrome requiring medical therapy.

1. Not currently treated with somatostatin receptor ligands agonists for at least 12 weeks prior to screening and actively symptomatic. This can include treatment-naïve subjects.
2. Subjects currently treated with lanreotide, octreotide long acting release, or short acting octreotide (subcutaneous or oral) who are currently symptomatically controlled
3. Evaluable documentation of locally advanced or metastatic histopathologically confirmed well-differentiated neuroendocrine tumor (NET). Tumors must be Grade 1 (Ki-67 index < 3%, or a mitotic count of < 2 mitoses per 10 high-power fields, if the Ki-67 index is not available) or Grade 2 (Ki-67 index 3-20%, or a mitotic count of 2-20 mitoses per 10 high-power fields, if the Ki-67 index is not available) per the World Health Organization neuroendocrine neoplasm classification (Rindi and Inzani, 2020). Grade 3 tumors are not eligible.
4. No significant disease progression as assessed by the Investigator within the last 6 months before initiation of study drug dosing.

Exclusion Criteria:

1. Diarrhea attributed to any condition(s) other than carcinoid syndrome.
2. Uncontrolled/severe diarrhea associated with significant volume contraction, dehydration, or hypotension.
3. Requires second line treatments (eg, telotristat) for control of carcinoid syndrome symptoms.
4. Treatment with specific NET tumor therapy <4 weeks before Screening (such as everolimus or sunitinib) or hepatic embolization, radiotherapy, peptide receptor radionuclide therapy (PRRT), and/or tumor debulking <12 weeks before Screening.
5. History of another primary malignancy <3 years prior to the date of first dose, except for adequately treated basal or squamous cell carcinoma of the skin, cancer of the breast or cervix in situ, previously treated or concurrent malignancy determined to be clinically stable and not requiring treatment.
6. Diabetes mellitus treated with insulin for less than 6 weeks prior to the study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (14):
  - Crinetics Study Site, Los Angeles, California
  - Crinetics Study Site, Newport Beach, California
  - Crinetics Study Site, Stanford, California
  - Crinetics Study Site, Miami, Florida
  - Crinetics Study Site, Iowa City, Iowa
  - Crinetics Study Site, Lexington, Kentucky
  - Crinetics Study Site, New Orleans, Louisiana
  - Crinetics Study Site, Boston, Massachusetts
  - Crinetics Study Site, Rochester, Minnesota
  - Crinetics Study Site, New York, New York
  - Crinetics Study Site, Stony Brook, New York
  - Crinetics Study Site, Cleveland, Ohio
  - Crinetics Study Site, Columbus, Ohio
  - Crinetics Study Site, Houston, Texas
- Argentina (2):
  - Crinetics Study Site, CABA, Buenos Aires
  - Crinetics Study Site, CABA
- Brazil (5):
  - Crinetics Study Site, Fortaleza, Ceará
  - Crinetics Study Site, Rio de Janeiro, Rio de Janeiro
  - Crinetics Study Site, Criciúma, Santa Catarina
  - Crinetics Study Site, São Paulo, São Paulo
  - Crinetics Study Site, Rio de Janeiro
- Crinetics Study Site, Toronto, Canada
- Mexico (2):
  - Crinetics Study Site, Mexico City, Cuauhtemoc
  - Crinetics Study Site, Querétaro City, Querétaro
- Peru (2):
  - Crinetics Study Site Peru #1, Lima
  - Crinetics Study Site Peru #2, Lima
- Poland (3):
  - Crinetics Study Site, Katowice
  - Crinetics Study Site, Warsaw
  - Crinetics Study Site, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In general, results are reported based on the dose assigned at randomization, regardless of the actual dose received.
Period: Overall Study
Arm/Group | 40 mg Paltusotine | 80 mg Paltusotine
Started | 18 | 18 (Dose adjustments could be made once at Week 2 or Week 4 if carcinoid syndrome symptoms met the criteria for short-acting octreotide rescue (dose increase), or if there was unacceptable tolerability of the randomized dose (dose decrease).)
Adverse Event | 1 | 1
Physician Decision | 0 | 3
Withdrawal by Subject | 0 | 1
Completed | 17 (Completed_RTP) | 13 (Completed_RTP)
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg Paltusotine | 80 mg Paltusotine | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Full Range); unit: years] | 58.6 [35 to 83] | 62.9 [41 to 78] | 60.8 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Europe | 1 | 1 | 2
  United States | 9 | 10 | 19
  South America | 8 | 7 | 15
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.057 (4.3181) | 28.609 (10.8261) | 28.833 (17.58)
Symptomatic Entry Criteria Met - n (%) [Count of Participants; unit: Participants]
  Bowel Movement Criteria Only | 6 | 8 | 14
  Flushing Criteria Only | 4 | 7 | 11
  Bowel Movement and Flushing Criteria | 8 | 3 | 11
Baseline Mean Daily Bowel Movements (/day) [Mean (Standard Deviation); unit: BMs per day] | 3.881 (2.0398) | 3.343 (1.3705) | 3.612 (1.7343)
Baseline Mean Daily Flushing Criteria Episode (/day) [Mean (Standard Deviation); unit: FE per day] | 2.325 (1.3219) | 2.413 (2.3313) | 2.369 (1.8683)
Duration Since Carcinoid Syndrome Diagnosis (Months) [Mean (Standard Deviation); unit: months] | 102.566 (82.0788) | 54.459 (37.1727) | 78.513 (67.3684)
Screening Group, n (%) [Count of Participants; unit: Participants]
  Not Currently on SRLs or Naïve to SRLs | 5 | 4 | 9
  Currently Treated with Lanreotide, Octreotide LAR, or Short-acting Octreotide | 13 | 14 | 27
Tumor Confirmation Method, n (%) [Count of Participants; unit: Participants]
  MRI | 9 | 5 | 14
  CT Scan | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Safety - Incidence of Treatment-emergent Adverse Events (TEAEs)
Description: Incidence of TEAEs, including serious TEAEs and TEAEs leading to discontinuation; change from baseline to the EOR in safety parameters: clinical laboratory tests, physical exam findings, vital signs, 12-lead ECG, and 24-hour continuous cardiac monitoring (only for subjects on 120 mg dose). In addition to all-cause mortality, deaths were categorized by primary cause (e.g., cardiovascular) based on medical adjudication. Events were coded using MedDRA and summarized by treatment group, system organ class, and preferred term.
  TEAEs were reported per randomized arm. There were 2 randomized arms (40 mg and 80 mg paltusotine, with up-or down-dose titration permitted for symptom control). Results are analyzed based on the initially assigned randomization arm, regardless of the actual dose received.
Time Frame: First dose of investigational medicine to End of Randomized Treatment Phase (8 weeks)
Population: Safety Analysis Set included all randomized participants receiving ≥1 dose. TEAEs (reported per randomized arm) are defined as AEs from first to last dose date (end of RTP, or early term), plus 28 days (Safety follow up). Dose changes at Weeks 2 or 4 were allowed for symptom control (increase) or poor tolerability (decrease). Results are provided by randomized arms (40 mg and 80 mg paltusotine).
Measure: Number; unit: participants
Arm/Group | 40 mg Paltusotine | 80 mg Paltusotine
Number analyzed (Participants) | 18 | 18
participants
  Treatment-Emergent Adverse Events (TEAE) | 16 | 15
  TEAE Related to CS Symptoms | 10 | 9
  Highest Severity of TEAE: Severe TEAE | 3 | 1
  Highest Severity of TEAE: Moderate TEAE | 6 | 7
  Highest Severity of TEAE: Mild TEAE | 7 | 7
  Serious TEAE | 2 | 2
  Treatment Related TEAE | 10 | 13
  Treatment Related Serious TEAE | 0 | 0
  TEAE Leading to Study Discontinuation | 1 | 1
  TEAE Leading to Actions Taken with Study Treatment: Dose Increased | 3 | 1
  TEAE Leading to Actions Taken with Study Treatment: Dose Decreased | 0 | 2
  Actions Taken with Study Treatment: Drug Withdrawn | 0 | 1
  Actions Taken with Study Treatment: Drug Interrupted | 3 | 2
  Actions Taken with Study Treatment: Dose Not Changed | 16 | 15
  Actions Taken with Study Treatment: Not Applicable | 2 | 4

2. Secondary Outcome: Pharmacokinetics (PK) of Paltusotine
Description: Steady state trough levels by dose and visit for Randomized Treatment Phase (RTP).
  The "Overall Number of Participants Analyzed" displayed at the top of the PK summary table represents the total number of participants who received each dose at any point during the trial, factoring in dose titrations. PK results are summarized by actual dose taken right before the time of sample collection, rather than by randomized dose. Participants may be included in different dose groups for different visits due to dose titration.
Time Frame: Measured at each visit (pre and post dose) up to Week 8 (i.e., End of Randomized Treatment Phase [EOR])
Population: The PK Analysis Set included all randomized participants with ≥1 paltusotine dose and ≥1 plasma measurement. Post-dose samples were taken 1-3 hrs after dosing, and steady-state troughs were assessed pre and post dose, through Week 8. Primary PK summaries were based on the RTP. Dose adjustments at Weeks 2 or 4 were allowed for symptom control (dose increase) or tolerability (dose decrease).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 40 mg Paltusotine: 40 mg paltusotine: Two 20 mg tablets QD
- 80 mg Paltusotine: 80 mg paltusotine: Four 20 mg tablets QD
- 120 mg Paltusotine: 120 mg paltusotine: Six 20 mg tablets QD
Arm/Group | 40 mg Paltusotine | 80 mg Paltusotine | 120 mg Paltusotine
Number analyzed (Participants) | 20 | 24 | 3
ng/mL
  WEEK 1 (POST-DOSE): number analyzed (Participants) | 18 | 17 | 0
  WEEK 1 (POST-DOSE) | 188 (80.8) | 360 (103.3) |
  WEEK 2 (PRE-DOSE): number analyzed (Participants) | 16 | 14 | 0
  WEEK 2 (PRE-DOSE) | 61.4 (153.5) | 193 (83.5) |
  WEEK 2 (POST-DOSE): number analyzed (Participants) | 14 | 18 | 1
  WEEK 2 (POST-DOSE) | 217 (90.5) | 473 (78.7) | 1240 (0.0)
  WEEK 4 (PRE-DOSE): number analyzed (Participants) | 16 | 17 | 1
  WEEK 4 (PRE-DOSE) | 68.2 (179.1) | 158 (74.7) | 218 (0.0)
  WEEK 4 (POST-DOSE): number analyzed (Participants) | 14 | 17 | 3
  WEEK 4 (POST-DOSE) | 209 (202.1) | 462 (82.7) | 545 (184.5)
  WEEK 6 (PRE-DOSE): number analyzed (Participants) | 11 | 17 | 3
  WEEK 6 (PRE-DOSE) | 57.8 (188.8) | 155 (63.1) | 146 (58.4)
  WEEK 6 (POST-DOSE): number analyzed (Participants) | 11 | 18 | 3
  WEEK 6 (POST-DOSE) | 261 (108.6) | 532 (89.4) | 474 (79.0)
  WEEK 8 - EOR (PRE-DOSE): number analyzed (Participants) | 10 | 16 | 2
  WEEK 8 - EOR (PRE-DOSE) | 63.3 (122.1) | 165 (44.5) | 201 (69.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 8 weeks of the RTP phase, and an EOS Visit was to occur to collect the safety data and other assessments, 28 days after last dose of study drug and was required for subjects who completed the study or early terminated. TEAE data were summarized from first dose date until last dose date (end of RTP or early term) plus 28 days (Safety follow up).
Description: AE results were reported based on the dose assigned at randomization (40 mg and 80 mg paltusotine), regardless of the actual dose received at the time of AE reporting. Dose changes at Weeks 2 or 4 were allowed for symptom control (increase) or poor tolerability (decrease).
Arm/Group | 40 mg Paltusotine | 80 mg Paltusotine
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/18
Serious Adverse Events (participants affected / at risk) | 2/18 | 2/18
Other Adverse Events (participants affected / at risk) | 16/18 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg Paltusotine (N=18) | 80 mg Paltusotine (N=18)
Cardiac failure (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Infections and infestations (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg Paltusotine (N=18) | 80 mg Paltusotine (N=18)
Diarrhoea (Gastrointestinal disorders) | 6 | 9
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Headache (Nervous system disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 2 | 5
Flushing (Vascular disorders) | 3 | 2
Fatigue (General disorders) | 2 | 2
Alanine aminotransferase increased (Investigations) | 0 | 3
Asthenia (General disorders) | 1 | 2
Amylase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 1
Blood creatinine increased (Investigations) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT05361668/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT05361668/SAP_001.pdf